CLINICAL TRIAL: NCT02866058
Title: Substantial Variability Between Traditional and Instrumental Variable Estimates of the Risk of Caesarean Section in Canada: a Population-based Cohort Study
Brief Title: Outcomes of Cesarean Section vs Vaginal Delivery: Instrumental Variable Adjusted Analysis
Status: Completed | Type: Observational
Sponsor: Memorial University of Newfoundland (Other)
Collaborators: Medical Research Foundation - Memorial University (Unknown)
Responsible Party: Principal Investigator, Kris Aubrey-Bassler, Director, Primary Healthcare Research Unit, Memorial University of Newfoundland
Other Study IDs: MRFCoxAwardAubrey2
Record Dates: First submitted 2016-08-04; First posted 2016-08-15 (Estimated); Last update posted 2016-08-15 (Estimated); Status verified 2016-08

CONDITIONS: Pregnancy Complications; Cesarean Section
MeSH Terms: conditions — Pregnancy Complications | interventions — Cesarean Section

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cesarean: Mothers delivered by cesarean section
  Interventions: Procedure: Cesarean Section
- Vaginal: Mothers delivered by vaginal delivery

INTERVENTIONS:
Procedure: Cesarean Section
  Groups: Cesarean

SUMMARY:
This study will examine the effect of cesarean section on perinatal mortality, using data provided by the Canadian Institute for Health Information.

DETAILED DESCRIPTION:
This study will examine administrative data provided by the Canadian Institute for Health Information (CIHI). Maternal obstetrical delivery and neonatal hospitalization records provided by CIHI will be linked before analysis. The primary outcome is in-hospital perinatal mortality. The data will be analyzed by traditional multi-variate logistic regression, and the results from this analysis will be compared to the results from instrumental variable adjusted regression using the Generalized Method of Moments. The instrumental variable is the rate of cesarean delivery among women living within the same hospital catchment area. All analyses will be adjusted for maternal, infant, delivery provider, and hospital factors, as well as for clustering at the level of the delivery hospital.

ELIGIBILITY:
Inclusion Criteria:

* Mothers living in Canada and their infants delivering within the study period at Canadian hospitals outside of the province of Quebec.

Exclusion Criteria:

* Maternal record not linkable to neonatal record.
* Multiple gestation.
* Birthweight < 500 gm.
* Gestational age at delivery < 20 weeks.
* Deliveries at hospitals with less than 20 cesarean deliveries during study period.
* Records with missing data for important covariates

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All obstetrical deliveries in Canada (except the province of Quebec) between April 1, 2006 and March 31, 2009
Sampling Method: Non-Probability Sample
Enrollment: 1703590 (Actual)
Dates: Start 2011-05; Primary Completion 2013-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Perinatal Mortality | up to 7 days
  Includes deaths at any age if infant continuously hospitalized (including transfers) in an acute care facility. Includes deaths up to 7 days of age if infant discharged from hospital then readmitted prior to 7 days of age.

CONTACTS AND LOCATIONS:
Overall Officials: Kris Aubrey-Bassler, MD, Principal Investigator — Memorial University

IPD SHARING:
Plan to Share IPD: No
The data provider does not allow sharing of investigator data, but data can be requested directly from them.